CLINICAL TRIAL: NCT06590454
Title: Therapeutic Intervention to Reverse Gastric Precancer
Brief Title: REVerse Intestinal Metaplasia in the Stomach (REVISE)
Acronym: REVISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Katherine Garman (Other)
Responsible Party: Sponsor-Investigator, Katherine Garman, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00115397; CA230416P2 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gastric Intestinal Metaplasia; Gastric Precancer
Keywords: Gastric Intestinal Metaplasia; Pyrvinium
MeSH Terms: interventions — pyrvinium

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial:
  Pyrvinium (n=16) Placebo (n=16)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pyrvinium (Active Comparator): Participants will receive Pyrvinium (2 mg/kg/day) by mouth once each day for a total of 14 days.
  Interventions: Drug: Pyrvinium
- Placebo (Placebo Comparator): Participants will receive placebo by mouth once each day for a total of 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyrvinium — Pyrvinium (2 mg/kg) per day for 14 days
  Arms: Pyrvinium
Drug: Placebo — Placebo for 14 days
  Arms: Placebo

SUMMARY:
This study is designed to test the use of Pyrvinium vs placebo as a treatment for gastric intestinal metaplasia with features associated with increased risk of cancer. Response will be determined by assessing the extent and quality of the gastric intestinal metaplasia before and after treatment.

A secondary aim will be to generate gastric organoids from patient-derived samples to test the effects of pyrvinium in vitro in patient-derived samples, and also to identify new drugs that may help reverse gastric intestinal metaplasia.

DETAILED DESCRIPTION:
The proposed study is an early Phase II Clinical Trial designed to generate additional data regarding safety and efficacy for the use of Pyrvinium, an FDA-approved drug no longer in active use. The study design includes enrollment in an observational cohort for a research-focused screening upper endoscopy to document the extent and type of gastric intestinal metaplasia in patients previously diagnosed with this condition using a standardized mapping protocol (as described below). This initial screening research endoscopy is needed as current clinical care is variable (due to lack of guidelines for mapping and surveillance). The investigators anticipate enrolling 60 participants in the observational cohort for intensive gastric mapping, and then of these 60 participants, 32 eligible participants (after determining eligibility based on presence of high-risk features of the gastric intestinal metaplasia with confirmed extensive gastric intestinal metaplasia) will be included in the randomized control trial to receive either Pyrvinium (n=16) or placebo (n=16).

Treatment is planned as followed:

2 weeks of Pyrvinium vs placebo (within 3 months of initial research endoscopy).

Following the initial endoscopy, participants will receive placebo or Pyrvinium (2 mg/kg/day) by mouth once each day for a total of 14 days. The drug (or placebo) will be verified and dispensed from the investigational drug pharmacy using an IND with attention to safety and blinding to research participants and clinical research staff. The drug and placebo will be administered as liquid suspensions. Medication diary logs will be used and participants will be asked to return bottles that contained the medication.

All participants will be advised to use sunblock and wear protective clothing due to potential for sun-sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (including men, women, and non-binary individuals) over age 18 with known GIM with at least one high-risk feature (extensive vs limited, incomplete or mixed-type GIM, family history of stomach cancer),
* Ability to provide informed consent,
* Evidence of prior but not active H. pylori infection

Exclusion Criteria:

* Active gastric cancer diagnosis,
* High-risk of bleeding complications due to anticoagulants or underlying medical condition,
* Pregnancy (which is a contraindication to non-emergent endoscopy due to anesthesia risks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of clinical biopsies with evidence of gastric intestinal metaplasia | Screening endoscopy (baseline) to the follow-up endoscopy (4-8 weeks)
  For the efficacy analysis, the investigators will primarily evaluate the change in the number of clinical biopsies with evidence of gastric intestinal metaplasia from the screening endoscopy to the follow-up endoscopy.

SECONDARY OUTCOMES:
Number of clinical biopsies with evidence of gastric intestinal metaplasia | 1 year
Number of clinical biopsies with complete gastric intestinal metaplasia | 1 year
Number of clinical biopsies with incomplete gastric intestinal metaplasia | 1 year
Number of clinical biopsies with presence of parietal cells (reversal of atrophy) | 1 year
Number of clinical biopsies with presence of inflammation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Garman, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No